CLINICAL TRIAL: NCT03709134
Title: Genomic Markers for Measuring Breast Cancer Response to Neoadjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Katarzyna Jerzak, Medical Oncologist & Associate Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 178-2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Cancer, Breast
Keywords: Circulating tumor cells; CTC; Circulating tumor DNA; ctDNA; Genomics; Transcriptomics
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Genomic Markers (CTC/ctDNA) — This is a non-interventional study.

SUMMARY:
The primary aim of the study is to identify genomic markers (circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), transcriptomic markers) as biomarkers of response to neoadjuvant chemotherapy (NAC) among patients with invasive breast cancer.

DETAILED DESCRIPTION:
The study aims to evaluate genetic markers (i.e. CTCs and ctDNA) in breast tumors to predict therapy response and metastatic risk. We aim to investigate genomic markers of treatment response and outcomes in breast cancer patients treated with neoadjuvant chemotherapy. The role of CTCs and ctDNA in predicting response to NAC will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give appropriate written informed consent prior to participation in the study.
2. Subjects must be women or men age 18+.
3. Subjects must be receiving neoadjuvant chemotherapy for breast cancer. All chemotherapy types and regimens are acceptable (systemic therapy will determined by the overseeing medical oncologist).
4. Biopsy-confirmed diagnosis of invasive breast cancer (i.e. ER+/-, PR+/-, HER2+/-).
5. Stage I-III disease according to the AJCC v7 criteria.

Exclusion Criteria:

1. Subjects with a past medical history of abnormalities, significant injury, or medical or surgical procedures (e.g. silicone/saline implants) involving either breast, exclusive of the lesion at issue.
2. Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study, such as significant anxiety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll women and men with a pathologically-confirmed diagnosis of invasive breast cancer that is stage I-III according to the AJCC v7 criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to 60 months
  Evaluating the degree of absence of residual cancer cells

SECONDARY OUTCOMES:
Time to distant breast cancer recurrence (months) | Up to 60 months
  Evaluating the time until a recurrence event has occurred in the breast.
Time to any recurrence (months) | Up to 60 months
  Evaluating the time until a local, regional, or distant recurrence event has occurred.
Time to death | Up to 60 months
  Evaluating time to cancer-related death

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna J Jerzak, MD, MSc, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided